CLINICAL TRIAL: NCT00716950
Title: Evaluation of Antihypertensive Activity of Valsartan and Amlodipine Compared to Losartan and Amlodipine Through Ambulatory Blood Pressure Monitoring in Moderate Hypertensive Patients in a Randomized, Controlled, Double-Blind Study
Brief Title: Valsartan and Amlodipine Compared to Losartan and Amlodipine in Hypertensive Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Responsible Party: Roberto Fogari/Full Professor of Internal Medicine, University of Pavia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UNIPV004DIM2008
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2008-07-17 (Estimated); Status verified 2008-07

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Valsartan; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): valsartan/amlodipine
  Interventions: Drug: valsartan/amlodpine
- 2 (Active Comparator): losartan/amlodpine
  Interventions: Drug: losartan/amlodpine

INTERVENTIONS:
Drug: valsartan/amlodpine — tablets; 160mg/5mg; od; 4 weeks
  Arms: 1
Drug: losartan/amlodpine — tablets; 100mg/5mg; od; 4 weeks
  Arms: 2

SUMMARY:
Hypertensive patients with moderate hypertension have a risk to develop cardiovascular events of 15-20% over a period of 10 years. It is important to reach quickly the advised target, but often this result can be obtained with a combination therapy. Some evidences demonstrate sartans and calcium channels blockers can be very useful and safe, but it is also important to verify which association can give side effects or give some pharmacokinetic interactions that can negatively influence the clinical combination efficacy.

ELIGIBILITY:
Inclusion Criteria:

* diastolic blood pressure in sitting position 100 to 109 mmHg and systolic blood pressure > 140 mmHg at the end of the selection period

Exclusion Criteria:

* type 2 diabetes mellitus
* heart failure
* AMI in the previous 6 months
* angina pectoris
* secondary hypertension
* malignant hypertension
* women child-bearing potential
* women who are pregnant and lactating
* suspected history of allergy to the sartans or calcium channels blockers

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
24 hours mean, determinated through ABPM; diastolic mean after 4 weeks of losartan 100mg/amlodipine 5mg and valsartan 160mg/amlodipine 5mg treatment | after 4 weeks

SECONDARY OUTCOMES:
24 hours systolic mean, determinated through ABPM; day systolic and diastolic mean determinated through ABPM; night systolic and diastolic mean determinated through ABPM | after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Fogari, MD, Study Chair — University of Pavia
Locations (1):
- Giuseppe Derosa, Pavia, Italy